CLINICAL TRIAL: NCT06515756
Title: The Effect of Three Different Bioceramic-Based Root Canal Sealers on Post-Operative Pain
Brief Title: Postoperative Pain Evaluation Of Novel Bioceramic-Based Root Canal Sealers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ali Turkyilmaz, Asisstant Professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 01.06.2023-07/06
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain, Acute
Keywords: Calcium-silicate,; Pain; Postobturation; Root canal sealer; Visual analog scale
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were blinded and were unaware of the specific treatment protocol. Participants were then randomly assigned to the four groups in a 1:1 ratio using a computer algorithm program (http:// randomizer.org)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All participates were divided into four experimantal groups according to the root canal sealers (Experimental): Participates were divided into four experimantal groups.
  Interventions: Other: Post operative pain assessment after root canal treatment
- Groups were divided into two subgroups to be applied on teeth with pulpitis and apical periodontitis (Experimental): Four different root canal sealer groups were divided into two subgroups to be applied on teeth with pulpitis and apical periodontitis. Although sealers were different, they was applied with the same technique.
  Interventions: Other: Post operative pain assessment after root canal treatment

INTERVENTIONS:
Other: Post operative pain assessment after root canal treatment — the sealer was administered to the root canal using the initial paper point and then uniformly distributed using a second paper point before removing any excess sealer with a third paper point. Once the sealer was applied, a single tapered gutta-percha cone was adjusted to fit the root canal. The coronal access cavities were restored with a composite resin material

SUMMARY:
Brief Summary: The purpose of this study was to evaluate the effect of MTA-Bioseal, GuttaFlow bioseal, and NeoSealer Flo calcium-silicate based root canal sealers on postobturation pain in teeth with asymptomatic irreversible pulpitis or chronic apical periodontitis undergoing single-visit root canal treatment.

The study tried to answer whether the type of sealer used altered the incidence and intensity of postobturation endodontic pain, whether pulp status affected the incidence and intensity of postobturation endodontic pain and whether there was no difference in analgesic intake by patients after a single-visit root canal treatment between the experimental groups.

DETAILED DESCRIPTION:
This prospective clinical study was reported pain levels experienced after obturation were similar for the different pulp statuses and root canal sealers tested. The participants with single-rooted teeth were included and divided into four groups according to the root canal sealer used. Then, the patients were divided into two subgroups according to pulp vitality. The postobturation pain scores were recorded after obturation on a visual analog scale (VAS) at 6, 12, 24, and 48 hours, and at 7 and 30 days. The level of pain experienced after obturation was similar for all root canal sealers in different pulp statuses. The results of the study showed that the bioceramic-based sealers tested can be used safely in clinical practice in terms of postobturation pain.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene,
* Not reporting pain before the appointment
* Asymptomatic irreversible pulpitis caused by deep carious lesions (vital cases),
* Asymptomatic primary apical periodontitis (non-vital cases).

Exclusion Criteria:

* Pregnancy,
* Autoimmune diseases,
* Uncontrolled diabetes,
* Smokers,
* Advanced periodontal disease (with 5 mm or more probing depth),
* Patients requiring endodontic treatment for more than one tooth,
* Unrestorable coronal destruction,
* Incomplete root formation, systemic,
* Allergic sensitivity to local anesthetic or NSAIDs.
* ASA II patient
* An analgesic or antibiotic intake the 7 days before the beginning of treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Change in pain from 6 th hours to 30 days between root canal sealers | 6, 24, and 72 hours and at 7 and 30 days
  All participants were asked to rate their perceived pain on the scale, with 0 indicating no pain and 10 indicating the highest possible pain. Pain levels were classified as none, mild (1 to 3), moderate (4 to 7), or severe (8 to 10).

SECONDARY OUTCOMES:
Change in pain from 6 th hours to 30 days between diffrernt pulp status | 6, 24, and 72 hours and at 7 and 30 days,
  All participants were asked to rate their perceived pain on the scale, with 0 indicating no pain and 10 indicating the highest possible pain. Pain levels were classified as none, mild (1 to 3), moderate (4 to 7), or severe (8 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Turkyilmaz, PhD, Study Director — Kirikkale University, Faculty of Dentistry
Locations (2):
- Turkey (Türkiye) (2):
  - Ali Turkyilmaz, Yahşihan, Kırıkkale
  - Ali Turkyilmaz, Kırıkkale

IPD SHARING:
Plan to Share IPD: No
The authors of the article could not reach a consensus on this issue.

REFERENCES:
- [Derived] Turkyilmaz A, Baris SD, Hancerliogullari D, Erdemir A. Postobturation Pain of three Novel Calcium Silicate-based sealers with asymptomatic irreversible pulpitis or necrotic pulp with chronic apical periodontitis: prospective clinical trial. BMC Oral Health. 2024 Nov 10;24(1):1366. doi: 10.1186/s12903-024-05161-1. PMID 39523312